CLINICAL TRIAL: NCT03698227
Title: Efficacy of Olaratumab and Rechallenge With Doxorubicin in Anthracycline Pretreated, Advanced Soft Tissue Sarcoma Patients. An Exploratory Phase-II Study
Brief Title: OlaReDo - Olaratumab and Rechallenge With Doxorubicin in Soft Tissue Sarcoma Patients
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Lack of efficacy on olaratumab
Sponsor: Institut für Klinische Krebsforschung IKF GmbH at Krankenhaus Nordwest (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OlaReDo_GISG-17
Record Dates: First submitted 2018-10-01; First posted 2018-10-05 (Actual); Last update posted 2020-07-15 (Actual); Status verified 2020-07

CONDITIONS: Advanced Soft Tissue Sarcoma
Keywords: Soft tissue sarcoma
MeSH Terms: conditions — Sarcoma | interventions — olaratumab; Pharmaceutical Preparations; Dexrazoxane; Doxorubicin

STUDY DESIGN:
Intervention Model Description: Olaratumab and doxorubicin rechallenge in anthracycline pretreated, advanced soft tissue sarcoma patients
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Study treatment (Experimental): * Olaratumab 20 mg/kg IV on day 1 and day 8 of cycle 1 and 15 mg/kg olaratumab IV on day 1 and day 8 of cycles 2-8.
  * Plus dexrazoxane at a dose equal to 10 times the doxorubicin dose (mg/m2) IV on day 1 of each 21 day cycle for 8 cycles
  * Plus doxorubicin 75 mg/m2 IV on day 1 of each 21 day cycle for 8 cycles
  * Beginning with cycle 9, olaratumab maintenance monotherapy at 15 mg/kg IV on day 1 and day 8 of each subsequent 21 day cycle
  Interventions: Drug: Olaratumab; Drug: Dexrazoxane; Drug: Doxorubicin

INTERVENTIONS:
Drug: Olaratumab — iv infusion
  Other Names: Study treatment
Drug: Dexrazoxane — iv infusion
  Other Names: Study treatment
Drug: Doxorubicin — iv infusion
  Other Names: Study treatment

SUMMARY:
This is an exploratory, prospective, open label, single arm, phase II-study for the evaluation of efficacy and feasibility (as determined by safety and tolerability) of olaratumab and doxorubicin rechallenge in anthracycline pretreated locally advanced (unresectable) or metastatic soft tissue sarcoma patients.

DETAILED DESCRIPTION:
Until now, rechallenge with anthracyclines in patients with metastatic STS which had a benefit from prior anthracycline containing therapy was never investigated in a prospective study.

Due to the very promising effect of olaratumab and doxorubicin in anthracycline-naïve patients and further taking into consideration the results of the retrospective anthracycline rechallenge study, there is a clear rationale to evaluate the effects of olaratumab and doxorubicin also in anthracycline pretreated patients by conducting a prospective clinical trial.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have histologically confirmed soft tissue sarcoma (STS) Note: Evidence of disease progression at study entry is required.
2. Treated in any order (neoadjuvant, adjuvant or for metastatic disease) with an anthracycline containing chemotherapy (The participant may have had any number of prior systemic cytotoxic therapies for advanced/metastatic disease. All previous anticancer treatments must be completed ≥ 3 weeks (21 days) prior to first dose of study drug.)
3. No progression on prior therapy with anthracyclines or within three months after stopping this therapy
4. Signed written informed consent
5. Men and women aged ≥ 18 years
6. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
7. Locally advanced (unresectable) or metastatic disease
8. Presence of measurable or non-measurable but evaluable disease as defined by the Response Evaluation Criteria in Solid Tumors (RECIST 1.1, Eisenhauer et al. 2009)
9. Adequate haematologic, organ, and coagulation function within 2 weeks (14 days) prior to enrollment:

   * Absolute neutrophil count (ANC) ≥ 1,500/mm3; G-CSF is not permitted within 2 weeks (14 days) prior to enrollment
   * Platelet count ≥ 100,000/mm3
   * Creatinine clearance ≥ 45 mL/min (calculated by using the Cockcroft-Gault formula (refer to study protocol Appendix 4)
   * Total bilirubin ≤ upper limit of normal (ULN). In patients with Gilbert's Syndrome, total bilirubin should be < 3 mg/dL
   * AST/ALT ≤ 3.0 x upper limit of normal (ULN); in case of liver involvement, AST/ALT ≤ 5.0 x are acceptable
   * Haemoglobin ≥ 9 g/dl. If haemoglobin <9 g/dl, blood transfusion is permitted. If haemoglobin cannot be enhanced to ≥ 9 g/dl, patient cannot be included into the study
   * International Normalized Ration (INR) ≤ 1.5 or prothrombin time (PT) ≤ 1.5 x ULN
   * Partial thromboplastin time (PTT or aPTT) ≤ 1.5 x ULN if not on anticoagulant therapy. For patients receiving anticoagulants, coagulation parameters within the intended or expected range for their therapeutic use are allowed. Patients must have no history of active bleeding (defined as within 14 days of first dose of study drug) or pathological condition that carries a high risk of bleeding (for example, tumor involving major vessels or known esophageal varices)
   * If routine urinalysis ≥2+ proteinuria, patient must have ≤1000 mg protein on a 24-hour urine, or urine protein/creatinine ratio ≤1 on spot urine
10. Left ventricular ejection fraction (LVEF) ≥50% assessed within 28 days prior to enrollment
11. Females of child-bearing potential must have a negative serum pregnancy test within 7 days prior to enrollment (refer to study protocol Appendix 3)
12. Females of child-bearing potential and males and must agree to use highly effective contraceptive precautions during the trial and up to 6 months following the last dose of study drug (refer to study protocol Appendix 3)
13. The participant has, in the opinion of the investigator, a life expectancy of at least 3 months

Exclusion Criteria:

1. Diagnosis of GIST or Kaposi sarcoma
2. Active central nervous system (CNS) or leptomeningeal metastasis (brain metastasis) at the time of enrollment. Participants with a history of a CNS metastasis previously treated with curative intent (for example, stereotactic radiation or surgery) that have not progressed on follow-up imaging, have been asymptomatic for at least 60 days and are not receiving systemic corticosteroids and/or anticonvulsants, are eligible. Participants with signs or symptoms of neurological compromise should have appropriate radiographic imaging performed before enrollment to rule out brain metastasis
3. Prior radiotherapy of the mediastinal/pericardial area or whole pelvis radiation
4. The participant has symptomatic congestive heart failure (CHF), or severe cardiac arrhythmia
5. The participant has unstable angina pectoris, angioplasty, cardiac stenting, or myocardial infarction within 6 months of enrollment
6. The participant has a QTcB interval calculated using Bazett's formula interval of >450 milliseconds (msec) for males and >470 msec for females on screening electrocardiogram (ECG)
7. Females who are pregnant or breastfeeding
8. Known allergy to any of the treatment components including a history of allergic reactions attributed to compounds of chemical or biological composition similar to olaratumab, dexrazoxane or doxorubicin
9. The participant has a known active fungal, bacterial, or viral infection including human immunodeficiency virus (HIV) or viral (A, B, or C) hepatitis (screening is not required)
10. Known history of active bleeding (defined as within 14 days of first dose of study drug) or pathological condition that carries a high risk of bleeding (for example, tumor involving major vessels or known esophageal varices)
11. History of another primary cancer, with the exception of i) curatively treated non-melanomatous skin cancer or ii) curatively treated cervical carcinoma in situ or iii) other primary non-haematologic malignancies or solid tumor treated with curative intent, no known active disease and no treatment administered during the last 3 years prior to enrollment
12. Electively planned or required major surgery during the course of the clinical trial
13. Any condition that, in the opinion of the investigator, would compromise the well-being of the participant or the study or prevent the participant from meeting or performing study requirements
14. On-treatment participation in another clinical study in the period 30 days prior to start of study treatment and during the study
15. Legal incapacity or limited legal capacity
16. Any condition that requires concomitant vaccination with yellow fever vaccine

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2018-11-12 (Actual); Primary Completion 2020-06-25 (Actual); Study Completion 2020-06-25 (Actual)

PRIMARY OUTCOMES:
Progression-free survival rate after 3 months (PFSR3), assessed by applying RECIST 1.1 | After 3 months treatment
  number of patients proven progression-free and alive after 3 months divided through the total number of patients in the all-treated-subjects population

SECONDARY OUTCOMES:
Progression free survival (PFS) | 6 months of Follow Up
  Time from the first dosing date of any study medication to the date of the first Objectively documented tumor progression, as determined by investigators (per RECIST v1.1), or death due to any cause.
Objective response rate (ORR) (i.e. CR or PR) | 6 months of Follow Up
  Number and percentage of participants with a best overall response (BOR) of complete response (CR) or partial response (PR)
Disease control rate (DCR) (i.e. CR, PR or SD) | 6 months of Follow Up
  Number and percentage of participants with complete response (CR) or partial response (PR) or stable disease (SD)
Overall survival (OS) | 6 months of Follow Up
  Time from date of the first dosing date of any study medication to the date of death (due to any cause)
Assessment of adverse events | During study conduct up to a maximum of 18 months (EOT)
  Type, incidence and severity of AEs, SAEs
Study therapy discontinuation rate due to cardiac toxicity | After treatment discontinuation up to a maximum of 18 months (EOS)
  Number of patients proven study therapy discontinuation due to cardiac toxicity (i.e. due to LVEF reduction by more than 20% or LVEF <45%) divided through the total number of patients in the all-treated-subjects population

CONTACTS AND LOCATIONS:
Overall Officials: Salah-Eddin Al-Batran, Prof. Dr., Study Director — Institut für Klinische Krebsforschung IKF GmbH at Krankenhaus Nordwest
Locations (4):
- Germany (4):
  - Helios Klinikum Bad Saarow, Bad Saarow
  - Helios Klinikum Berlin-Buch Klinik für Onkologie und Palliativmedizin, Berlin
  - Charité Universitätsmedizin Berlin Medizinische Klinik m. S. Hämatologie, Onkologie und Tumorimmunologie Campus Virchow Kliniken, Berlin
  - Medizinische Fakultät Carl Gustav Carus Medizinische Klinik I Internistische Onkologie, Dresden

IPD SHARING:
Plan to Share IPD: No
No IPD will be shared